CLINICAL TRIAL: NCT05907148
Title: Effects of Sensory Integration Training on Balance and Confidence in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-367-04-2023
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Sensory Integration Training; Berg Balance Scale; Balance; Activities-Specific Balance Confidence Scale
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Physical therapy along with Coordination exercises (Active Comparator): The Control group training will consist of active joint mobilization, muscle stretching, motor coordination exercises and additionally will receive 30-minute general balance training. Active joint mobilization will be carried out with the patient in the supine, prone (if possible), or sitting positions. Muscle stretching will be carried out mainly in the supine, prone (if possible), and standing positions. Motor coordination exercises will be carried out in a supine position, sitting and standing positions.
  Interventions: Other: Routine physical therapy; Other: General coordination exercise
- sensory Integration training group along with Routine physical therapy (Experimental): experimental group training will consist of active joint mobilization, muscle stretching, motor coordination exercises and additionally 30 minutes of sensory integration therapy.
  Interventions: Other: Sensory integration training; Other: Routine physical therapy

INTERVENTIONS:
Other: Sensory integration training — Sitting position:
  1. Sit in a chair without a backrest while the feet on firm surface. without backrest while the feet on soft surface.
  2. Sit on a ball while the feet on firm surface. while feet on soft surface.
  3. Sit in a chair without a backrest with the feet on firm surface and perform sit-to-stand motion.
     without a backrest with the feet on soft surface and perform sit-to-stand motion.
  4. Sit on a ball with the feet on the firm surface and perform sit-to-stand motion. with the feet on the soft surface and perform sit-to-stand motion.
  5. Perform bipedal standing on a firm surface. on a soft surface.
  6. Perform a semi-tandem stance on firm surface. on soft surface.
  7. Walk forward on firm surface. on soft surface.
  8. Walk forward on firm surface, cross obstacle, and continue to walk.
  9. Walk forward on the soft surface, cross obstacle, and continue to walk.
  Arms: sensory Integration training group along with Routine physical therapy
Other: Routine physical therapy — It consist of active joint mobilization, muscle stretching, motor coordination exercises and general balance training
  Other Names: consist of active joint mobilization, muscle stretching, motor coordination exercises and additionally will receive 30-minute general balance training.
Other: General coordination exercise — In supine lying:
  1. Patients are told to place heel of one leg on shin or knee of the other leg,
  2. Patient bends one leg and extends the other leg like bicycling motion.
  3. Flexing one leg while extending other leg
  4. Flexing and extending of one leg while abduction and adduction of other leg.
  In sitting:
  1. Patient performs marching without backrest or back support,
  2. Patient reaches forward and sideways with arms
  3. Rotation of trunk with physioball in hand without back support.
  4. Patient reaches with legs to marked point in sitting.
  In standing:
  Patient performs 10 repetitions of
  1. Clock Reach
  2. Side Leg Raises
  3. Leg Swings and
  4. Ball catch and throw
  Arms: Routine Physical therapy along with Coordination exercises

SUMMARY:
The Objective of this research was to study the effectiveness of sensory integration training on balance and confidence in patients with Parkinson's disease.

Null Hypothesis:

Sensory integration training and conventional balance training have no significant difference in improving balance and confidence of patients with Parkinson's disease.

Alternative Hypothesis:

Sensory integration training and conventional balance training have a significant difference in improving balance and confidence in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The study design will be randomized controlled clinical trial. Patients who fulfill the inclusion criteria will be identified by individual physiotherapist and will be enrolled for particular study. A sample size of 46 patients will be taken in this study by expecting a mean change 10.42 using 80% power of study and 95% level of significance and 20% dropout will also be included. So each group contains 23 participants.

The study will be single blinded. The outcome assessor will be unaware of the treatment given to both groups. Sample will be collected through simple random sampling technique, and randomization sequencing will be generated with help of lottery. After selection the sample patients will be divided into two groups, allocation concealment will be ensured by using sealed envelopes. Group A will be given conventional balance training along with routine physical therapy without sensory integration and Group B will be given sensory integration physical therapy along with routine physical therapy. Group A will be called control group and Group B will be called experimental group. Every patient has to pick up an envelope which will be placed in patient's file which later will be opened by the researcher who will provide patient treatment accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed by a neurologist with Parkinson's disease.
* Patients having BBS score between 21-40
* At least 6 months post neurological Sensory/Motor deficit patient.
* Age between 30 -65 years.
* Ability to maintain standing position without aids for at least 5 minutes.
* Normal vision
* No severe systemic disorders
* An ability to understand and perform the test

Exclusion Criteria:

* Patients with other existing neuromuscular disorders or medical conditions that substantially influences their gait and balance performance
* Neuropathy patients
* Vestibular disorders, paroxysmal vertigo.
* Presence of orthopedic conditions involving the lower limbs.
* Patients with psychiatric disorders.
* Pregnant patients.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS): | the change in the ability to balance in individual at baseline, 6th and 12th week
  The BBS is a 14-item validated scale that assesses static and dynamic Balance disorders in individuals with Parkinson's disease (score range, 0-56; higher=better performance). The items explore the ability to sit, stand, lean, turn, and maintain the upright position on one leg. Performance of these tasks depends on central integration processes to select specific response strategies which, in turn, depend on the characteristics of external postural displacement and goals
Activities-specific Balance Confidence Scale (ABC): | the change in the ability to balance in individual at baseline, 6th and 12th week
  This validated and reliable self-reported measure evaluates the patient's perceived level of balance confidence in performing various ambulatory activities without falling or experiencing a sense of instability. The overall score is calculated by adding the item scores and then dividing by the total number of items (score range, 0-100 points per activity; higher=more confident.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - ganga Raam Hopital, Lahore, Punjab Province
  - the Univerity of Lahore Teaching hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided